CLINICAL TRIAL: NCT06042608
Title: Effect of Adding an Intercostobrachial Nerve Block to an Interscalene Block on Postoperative Pain After Total Shoulder Arthroplasty
Brief Title: Evaluating Intercostobrachial Nerve Block's Effect on Pain Control After Shoulder Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Lisa Gu, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU-2023-0163
Record Dates: First submitted 2023-09-06; First posted 2023-09-18 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Postoperative Pain, Acute; Shoulder Pain
MeSH Terms: conditions — Pain, Postoperative; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active intercostobrachial nerve block (Active Comparator): Patient will receive local anesthetic injected around their intercostobrachial nerve in the axilla (armpit). They will still receive an active interscalene nerve block (gold standard) that helps with the rest of the shoulder pain.
  Interventions: Procedure: intercostobrachial nerve block
- Sham intercostobrachial nerve block (Placebo Comparator): Patient will receive saline injected around their intercostobrachial nerve in the axilla (armpit). This is a sham intercostobrachial nerve block because saline is not an active medication. They will still receive an active interscalene nerve block (gold standard) that helps with the rest of the shoulder pain.
  Interventions: Procedure: intercostobrachial nerve block

INTERVENTIONS:
Procedure: intercostobrachial nerve block — injection of local anesthetic to target the intercostobrachial nerve in the axilla

SUMMARY:
Interscalene blocks are frequently performed to decrease postoperative pain after shoulder surgeries and are considered the gold standard for pain control after this type of surgery. Some patients report pain in the axilla (armpit) following shoulder replacement surgeries. Sensation in the axilla is supplied by nerves not covered by the interscalene block. Sensation in the axilla can be decreased by performing an intercostobrachial nerve block. This study aims to study whether adding an intercostobrachial nerve block to the interscalene block decreases recovery room stay time, opioid pain medication requirement, and postoperative pain scores.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18-80 years old
* Adult patient's BMI <= 35
* Individuals presenting for primary total shoulder arthroplasty or reverse total shoulder arthroplasty
* Anticipated discharge home same day of surgery
* Patient is able to provide informed consent to participate in the study.

Exclusion Criteria:

* Patient presenting for revision shoulder surgery
* Allergy to amide local anesthetic, liposomal bupivacaine or other medication involving liposomal formulation
* Preexisting neurological deficits involving or potentially involving the ipsilateral brachial plexus
* Preexisting contralateral vocal fold paralysis or recurrent laryngeal paralysis
* Psychiatric or cognitive disorders that could interfere with perioperative evaluation including drug or alcohol abuse
* Chronic pain conditions
* Preoperative opioid use
* Moderate to severe pulmonary disease
* Moderate to severe sleep apnea
* Planned postoperative admission.
* Unplanned postoperative admission
* Any contraindication to interscalene or intercostobrachial nerve block including any local disorder of the skin where blockade is to be performed which would prevent safe performance of the block
* Any coagulation abnormality which would be a contraindication for block placement
* Preoperative chronic renal dysfunction requiring renal replacement therapy or CrCl < 60
* Sulfa allergy (or other reason patient cannot receive celecoxib)
* Allergy or intolerance to any medication in the protocol
* Body mass index >35
* Pregnancy
* Incarceration
* ASA classification greater than 3
* Inability to provide informed consent
* Refusal to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
time spent in PACU (recovery room) | 0-2 hours after surgery
amount of opioid pain medications required to control postoperative pain | 0-3 days after surgery

SECONDARY OUTCOMES:
pain scores (1-10 out of 10) | 0-3 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Farzin Ahmed, Study Director — farzin.ahmed@utsouthwestern.edu
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No